CLINICAL TRIAL: NCT05379738
Title: APALLO : Post Allogeneic Stem Cell Transplantation Adapted Physical Activity for Patient With Hematological Malignancies
Brief Title: Impact of Adapted Physical Activity on Patient's Recovery Following Allogeneic Stem Cell Transplantation for Hematological Malignancy
Acronym: APALLO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 21-PP-12
Record Dates: First submitted 2022-05-09; First posted 2022-05-18 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Haematological Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- adapted physical activity (Experimental): 6 sessions of physical activity
  Interventions: Other: 6 sessions of adapted physical activity after stem cell transplant

INTERVENTIONS:
Other: 6 sessions of adapted physical activity after stem cell transplant — physical assessement before and after stem cell transplant:
  * weight loss
  * brachial muscle circumference
  * grip strength evaluation
  * short physical battery test
  psychometric assessment before and after stem cell transplant:
  * quality of life questionary
  * physical activities questionary

SUMMARY:
It is a study about adaptated physical activity for patients receiving a stem cell transplantation. They will benefit of 6 adaptated individuals lessons at home between 1 month and 3 months after stem cell transplantation. The study's goal is to observe if adaptated activity has an positive impact on weight loss and on life quality.

ELIGIBILITY:
Inclusion criteria :

* Patient aged 18 or more
* Patient with social security
* Patient who accept the study and sign the consent form
* Patient programmed for an allogenic stem cell transplantation

Non inclusion criteria :

* Patients with a guardianship
* Patients with a significant additional physic or mental disease

Exclusion criteria

* Patients who did not receive an allogeniac stem cell transplantation
* Patients still hospitalized between day 30 and day 100 after stem cell transplantation
* Patients who finally refuses the study
* Patients who develop a physical or mental incapacity to practice physical activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-06-10 (Actual); Primary Completion 2026-12-10 (Estimated); Study Completion 2028-04-10 (Estimated)

PRIMARY OUTCOMES:
weight loss | before stem cell transplantation, 1 month , 3 months, 1 year after stem cell transplantation
  Body weight n in kilograms
weight loss | before stem cell transplantation, 1 month , 3 months, 1 year after stem cell transplantation
  Calculation of the percent of body weight loss between the " before stem cell transplantation evaluation " and each evaluation after stem cell transplantation and after adaptated physical activity sessions.

SECONDARY OUTCOMES:
patient's ability to attend the classes | 3 months after stem cell transplantation
  number of adaptated physical activity lessons attended by each patient after stem cell transplantation, calculation of feasibility
body mass index | before stem cell transplantation, 1 month , 3 months, 1 year after stem cell transplantation
  Measure of weight and height to evaluate the nutriotional status of a patient
brachial muscle circumference | before stem cell transplantation , 1 month , 3 months, 1 year after stem cell transplantation
  evaluation in centimeters of the brachial circumference to evaluate the evolution of the muscle circumference after stem cell transplantation and adaptated physical activity compared to the evaluation before stem cell transplantation. Using a measuring tape
grip strength evaluation | before stem cell transplantation , 1 month , 3 months, 1 year after stem cell transplantation
  it is a measure of muscular strength
short physical battery test | before stem cell transplantation , 1 month , 3 months, 1 year after stem cell transplantation
  it is a series of 3 physical tests to evaluate mobility the first test is a balance test (4 points), the second test is an evaluation of a walking speed (4 points) and the third test is a Chair rise test (4 points) The global test is on 12 points (12 is the better score)
Quality of Life Questionary C30 (QLQ-C30) | before stem cell transplantation , 1 month , 3 months, 1 year after stem cell transplantation
  it is a score to evaluate the quality of life of patients facing illness The subscales scores are transformed to a 0 to 100 scale, with higher score on functionnal scales indicating better function and higher scores on sumptom scales indicating worse symptoms
in house developped physical activities questionary | before stem cell transplantation , 1 month , 3 months, 1 year after stem cell transplantation
  it is a questionnary created especially for this study to evaluate on each step the capacity of each patient to maintain physical activities (social activities, autonomy at home for cooking and hygiene care, autonomy for transport to go to hospital appointments)

CONTACTS AND LOCATIONS:
Overall Officials: SOLDATI Alizée, Principal Investigator — CHU NICE, hopital ARCHET 1, hématologie
Locations (1):
- CHU NICE, hopital ARCHET 1, hématologie, Nice, France